CLINICAL TRIAL: NCT02182401
Title: An Open-label, Fixed Sequence Phase I Study in Healthy Male Volunteers to Assess Sequentially the Effects of Multiple Doses of BI 207127 NA, BI 201335 NA Followed by the Combination of BI 207127 NA and BI 201335 NA, on the Single Dose Pharmacokinetics of Midazolam and Tolbutamide and on the Systemic Exposure of BI 207127 NA and BI 201335 NA
Brief Title: Multiple Doses of BI 207127 NA, BI 201335 NA Followed by the Combination of BI 207127 NA and BI 201335 NA in Healthy Male Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1241.18
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Tolbutamide

ARMS (1):
- BI 207127 NA (Experimental): fixed sequence
  Interventions: Drug: BI 207127 NA; Drug: BI 201335 NA; Drug: Midazolam; Drug: Tolbutamide

INTERVENTIONS:
Drug: BI 207127 NA — Days 3-8 and days 25-30
Drug: BI 201335 NA — Days 15-30
Drug: Midazolam — Days 1, 7, 23 and 29
Drug: Tolbutamide — Days 1, 7, 23 and 29

SUMMARY:
Study to investigate the pharmacokinetic drug-drug interaction potential of BI 207127 NA and BI 201335 NA on each other at steady-state and to quantify the effect of BI 207127 NA, and BI 207127 NA combined with BI 201335 NA, on the activity of CYP 2C9 and CYP 3A4 using the probe substrates tolbutamide (CYP 2C9) and midazolam (CYP 3A4).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males (caucasian)
* Age ranging ≥ 21 and ≤ 50 years
* Body mass index (BMI) ≥ 19 and ≤ 29.9 kg/m2
* Willing to complete all study-related activities
* Volunteers give their written informed consent prior to admission to the study

Exclusion criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of photosensitivity or recurrent rash
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the trial or during the trial
* vulnerable subjects (that is persons kept in detention)
* exclusion of contraindications or hypersensitivity to midazolam and / or tolbutamide
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication and/or related drugs of these classes
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF, or QTcB interval >450 ms)
* Homozygous carriers of the UGT1A1 (uridine diphosphate glucuronosyltransferase 1A1) enzyme polymorphism *28 and *60

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Steady-state Cmax (Maximum measured concentration of the analyte in plasma) | up to day 31
Steady-state AUC (Area under concentration-time curve) | up to day 31

SECONDARY OUTCOMES:
Cmax for several time points | up to day 31
Tmax (Time from dosing to the maximum measured concentration of the analyte in plasma) | up to day 31
Cx for several time points | up to day 31
AUC for several time points | up to day 31
CL/F (Total apparent clearance of the analyte in plasma following extravascular administration) for several time points | up to day 31
V/F (Apparent volume of distribution during following an extravascular dose) for several time points | up to day 31
t1/2 (Terminal half-life of the analyte in plasma) | up to day 31
Cavg0-24 | up to day 31
Ratio for Cmax,Met at several time points | up to day 31
Ratio for AUC at several time points | up to day 31
Tlast,N | up to day 31
Ae (amount of analyte eliminated in urine for different time points) | up to day 29
CLR (renal clearance of the analyte for different time points) | up to day 29
fe (fraction of analyte eliminated in urine for different time points) | up to day 29
Number of patients with adverse events | up to 66 days
Assessment of tolerability on a 4-pointe scale by investigator | within 14 days after last drug administration